CLINICAL TRIAL: NCT03674814
Title: A Phase I Trial of Enzalutamide Plus the Glucocorticoid Receptor Antagonist CORT-125134 (Relacorilant) for Patients With Metastatic Castration Resistant Prostate Cancer (CRPC)
Brief Title: Study of Drug 1 (Enzalutamide) Plus Drug 2 (Relacorilant) for Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Corcept Therapeutics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-0152; P50CA180995 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-09-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; Enzalutamide; Relacorilant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; relacorilant

STUDY DESIGN:
Intervention Model Description: Patients will be sequentially enrolled to increasing dose escalation cohorts based on safety and PK.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Level (Experimental): Relacorilant will be given at a dose once daily. Enzalutamide will be given at a dose once daily.
  Interventions: Drug: Enzalutamide; Drug: Relacorilant

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide will be taken by mouth at assigned dose. Enzalutamide will be obtained as standard of care prescription (not provided by study).
  Other Names: Xtandi(R)
Drug: Relacorilant — Relacorilant will be taken by mouth at assigned dose. Relacorilant will be provided by the study.
  Other Names: CORT-125134

SUMMARY:
The study is an open-label Phase 1 study of the combination of relacorilant with enzalutamide in patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The study is an open-label Phase 1 study of the combination of relacorilant with enzalutamide in patients with metastatic castration resistant prostate cancer (mCRPC). Patients will be enrolled in 6 patient cohorts with a 6+3 design and a 28 day DLT period. Doses of relacorilant, enzalutamide will be adjusted based on safety and pharmacokinetics (PK). Once a safe dose with appropriate drug levels (PK) has been established, the cohort will be expanded to a total of 12 patients to refine safety and PK at the recommended phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate cancer with documented metastatic disease
2. Evidence of castrate testosterone level <50ng/dl (or surgical castration)
3. Evidence of disease progression:

   * 2 or more new lesions on bone scan or
   * Progressive disease on CT/MRI according to Response Evaluation Criteria in Solid Tumors 1.1 criteria or
   * Rising Prostate Specific Antigen (PSA): PSA evidence for progressive prostate cancer consists of a minimum PSA level of at least 2 ng/ml, which has subsequently risen on at least 2 successive occasions, at least 2 weeks apart.
4. Prior treatment with at least one line of potent androgen receptor signaling inhibitor (e.g. abiraterone, enzalutamide, apalutamide) in either castration-sensitive or castration-resistant setting.
5. Any prior therapy for castrate disease is acceptable except prior GR antagonist treatment (e.g. mifepristone or relacorilant).
6. Any other radiotherapy or radionuclide require 28-day washout prior to first dose of study drug.
7. Denosumab or zoledronic acid are allowed.
8. ECOG performance status ≤ 2.
9. Patients must have normal hepatic function as defined below:

   * Total bilirubin </=1.5 x the upper limit of normal
   * AST(SGOT)/ALT(SGPT) </=2.5 X institutional upper limit of normal
   * Albumin >/=3.0 g/dL
10. Patients must have normal bone marrow function as defined below:

    * Platelet count (plt) >/= 80,000 /microliter
    * Hemoglobin (Hgb) >/= 9 g/dL
    * Absolute neutrophil count (ANC) >/= 1500
11. Patients must have normal renal function as defined below:

    * GFR >/= 30 mL/min
12. Ability to understand and the willingness to sign a written informed consent document.
13. Patients with active Diabetes Mellitus on glucose lowering medications are eligible provided they agree to and are able to self-monitor daily blood glucose levels due to potential risk of lowering glucose levels on relacorilant.
14. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 3 months after final study drug administration. Two acceptable methods of birth control thus include the following:

    * Condom (barrier method of contraception); AND
    * One of the following is required:

      1. Established use of oral, or injected or implanted hormonal method of contraception by the female partner;
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner;
      3. Additional barrier method: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository by the female partner;
      4. Tubal ligation in the female partner;
      5. Vasectomy or other procedure resulting in infertility (e.g., bilateral orchiectomy), for more than 6 months.

Exclusion Criteria:

1. Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart), or any herbal product known to decrease PSA levels (e.g., saw palmetto and PC-SPES), or any systemic corticosteroid within 2 weeks prior to first dose of study drug.

   a.Patients who have been on systemic corticosteroids with prednisone equivalent of 10mg or greater for greater than 3 months immediately prior to participation in this study must have documented ability to tolerate cessation of corticosteroids prior to enrollment.
2. Inability to swallow capsules or known gastrointestinal malabsorption.
3. Evidence of visceral disease on imaging in a patient who is an appropriate candidate for cytotoxic chemotherapy (docetaxel or cabazitaxel).
4. History of other malignancies, with the exception of: adequately treated non-melanoma skin cancer, adequately treated superficial bladder cancer, stage 1 or 2 malignancies who are without evidence of disease, or other cancers curatively treated with no evidence of disease for > 5 years from enrollment.
5. Blood pressure that is not controlled despite > 2 oral agents (SBP >160 and DBP >90 documented during the screening period with no subsequent blood pressure readings >160/100).
6. History of seizure disorder or active use of anticonvulsants. Medications used to treat neuropathic pain such as gabapentin or pregabalin are allowed.
7. Documented history of or current brain metastases due to seizure risk
8. Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled.
9. Active psychiatric illness/social situations that would limit compliance with protocol requirements.
10. NYHA class II, NYHA class III, or IV congestive heart failure (any symptomatic heart failure).
11. Concurrent therapy with strong inhibitors or inducers of CYP3A4 or CYP2C8 (See Section 9.12below for list of strong inhibitor or inducers) due to concerning possible drug-drug interactions
12. Presence of concurrent medical conditions requiring systemic glucocorticoids for immunosuppression (e.g. Autoimmune diseases, organ transplantation) that is active and has required glucocorticoids in the last 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 28 days after start of dosing
Change in steady-state (C-trough) enzalutamide caused by relacorilant | 28 days after start of dosing

SECONDARY OUTCOMES:
Preliminary anti-cancer activity of relacorilant as measured by prostate specific antigen levels per response evaluation criteria in solid tumors | 12 weeks after initial start of combination dosing
Preliminary anti-cancer activity of relacorilant as measured by tumor response per response evaluation criteria in solid tumors | 12 weeks after initial start of combination dosing
Assess steady state relacorilant drug levels when given with enzalutamide | 28 days after start of dosing
Assess steady state enzalutamide drug levels when given with relacorilant | 28 days after start of dosing
Radiographic progression free survival (PFS) of the combination | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, MD, Principal Investigator — University of Chicago
Locations (1):
- University Of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Serritella AV, Shevrin D, Heath EI, Wade JL, Martinez E, Anderson A, Schonhoft J, Chu YL, Karrison T, Stadler WM, Szmulewitz RZ. Phase I/II Trial of Enzalutamide and Mifepristone, a Glucocorticoid Receptor Antagonist, for Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2022 Apr 14;28(8):1549-1559. doi: 10.1158/1078-0432.CCR-21-4049. PMID 35110415